CLINICAL TRIAL: NCT05455086
Title: Free-Base Nicotine or Nicotine Salt e-Liquids in Current E-Cigarette Smokers, PeloPET
Brief Title: Free-Base Nicotine or Nicotine Salt e-Liquids in Current E-Cigarette Smokers, PeloPET Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Theodore Wagener, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: OSU-21069; NCI-2021-05882 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-09-20; First posted 2022-07-13 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Cigarette Smoking-Related Carcinoma
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (pronated e-liquid, unprotonated e-liquid (Experimental): VISIT 2: Patients receive 1 puff of tobacco flavored or unflavored protonated e-liquid and undergo 0-15 min head and 5 min chest PET?CT and then 0-15 min chest and 5 min head PET/CT. About 2 hours post initial PET/CT, patients receive a second puff of tobacco flavored or unflavored protonated e-liquid and undergo 0-15 min chest and 5 min head PET/CT and then 0-15 min head and 5 min chest PET/CT.
  VISIT 3: Patients receive 1 puff of tobacco flavored or unflavored unprotonated e-liquid and undergo 0-15 min head and 5 min chest PET/CT and then 0-15 min chest and 5 min head PET/CT. About 2 hours post initial PET/CT, patients receive a second puff of tobacco flavored or unflavored protonated e-liquid and undergo 0-15 min chest and 5 min head PET/CT and then 0-15 min head and 5 min chest
  Interventions: Behavioral: Cigarette Smoking; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Other: Questionnaire Administration
- Arm II (unprotonated e-liquid, protonated e-liquid (Active Comparator): VISIT 2: Patients receive 1 puff of tobacco flavored or unflavored unprotonated e-liquid and undergo 0-15 min head and 5 min chest PET/CT and then 0-15 min chest and 5 min head PET/CT. About 2 hours post initial PET/CT, patients receive a second puff of tobacco flavored or unflavored unprotonated e-liquid and undergo 0-15 min chest and 5 min head PET/CT and then 0-15 min head and 5 min chest.
  VISIT 3: Patients receive 1 puff of tobacco flavored or unflavored protonated e-liquid and undergo 0-15 min head and 5 min chest PET/CT and then 0-15 min chest and 5 min head PET/CT. About 2 hours post initial PET/CT, patients receive a second puff of tobacco flavored or unflavored protonated e-liquid and undergo 0-15 min chest and 5 min head PET/CT and then 0-15 min head and 5 min chest PET/CT.
  Interventions: Behavioral: Cigarette Smoking; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Cigarette Smoking — Receive 1 puff of tobacco flavored protonated e-liquid
Behavioral: Cigarette Smoking — Receive 1 puff of unflavored protonated e-liquid
Behavioral: Cigarette Smoking — Receive 1 puff of tobacco flavored unprotonated cigarette
Behavioral: Cigarette Smoking — Receive 1 puff of unfavored unprotonated cigarette
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies the effect of free-base compared with nicotine salt based e-liquids on electronic cigarette (EC) puffing behavior, abuse liability, and deposition and absorption of nicotine in the respiratory tract and rate of uptake in the brain in current EC smokers. The results from this study may provide much needed scientific information to public health officials and regulators.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine the influence of nicotine form on puffing behavior and abuse liability.

II. To evaluate the influence of nicotine form and concentration on nicotine distribution in the brain and respiratory tract.

OUTLINE:

VISIT 1: Patients sample 4-liquids to determine whether they can vape the unflavored e-liquid without coughing

Patients are randomized to 1 of 2 arms.

ARM I:

VISIT 2: Patients receive 1 puff of tobacco flavored or unflavored protonated e-liquid and undergo 0-15 minutes (min) head and 5 min chest positron emission tomography (PET)/computed tomography (CT) and then 0-15 min chest and 5 min head PET/CT. About 2 hours post initial PET/CT, patients receive a second puff of tobacco flavored or unflavored protonated e-liquid and undergo 0-15 min chest and 5 min head PET/CT and then 0-15 min head and 5 min chest PET/CT.

VISIT 3: Patients receive 1 puff of tobacco flavored or unflavored unprotonated e-liquid and undergo 0-15 min head and 5 min chest PET/CT and then 0-15 min chest and 5 min head PET/CT. About 2 hours post initial PET/CT, patients receive a second puff of tobacco flavored or unflavored unprotonated e-liquid and undergo 0-15 min chest and 5 min head PET/CT and then 0-15 min head and 5 min chest

ARM II:

VISIT 2: Patients receive 1 puff of tobacco flavored or unflavored unprotonated e-liquid and undergo 0-15 min head and 5 min chest PET/CT and then 0-15 min chest and 5 min head PET/CT. About 2 hours post initial PET/CT, patients receive a second puff of tobacco flavored or unflavored unprotonated e-liquid and undergo 0-15 min chest and 5 min head PET/CT and then 0-15 min head and 5 min chest.

VISIT 3: Patients receive 1 puff of tobacco flavored or unflavored protonated e-liquid and undergo 0-15 min head and 5 min chest PET/CT and then 0-15 min chest and 5 min head PET/CT. About 2 hours post initial PET/CT, patients receive a second puff of tobacco flavored or unflavored protonated e-liquid and undergo 0-15 min chest and 5 min head PET/CT and then 0-15 min head and 5 min chest PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* A current exclusive e-cigarette user (>= 1 vaping bout per day) for at least the past 6 months (confirmed by NicAlert saliva testing strip)
* Between 21-50 years old
* Willing to provide informed consent and abstain from all tobacco and nicotine use for at least 12 hours prior to visits 2 and 3
* Willing to participate in 3 laboratory visits
* Read and speak English
* If utilizing study provided rideshare services, will need to live within 20 miles of Wake Forest University

Exclusion Criteria:

* Self-reported diagnosis of lung disease including asthma, cystic fibrosis, or chronic obstructive pulmonary disease
* Unstable or significant psychiatric conditions (past and stable conditions will be allowed)
* History of cardiac event or distress within the past 3 months
* Currently pregnant (as indicated by urine pregnancy test at the start of each laboratory visit), planning to become pregnant, or breastfeeding (women only)
* Use of other tobacco products (e.g., cigarette, cigar, etc.) > 5 days in the past month
* Currently engaging in a tobacco product cessation attempt

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore L Wagener, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant was consented and enrolled in the study but found to be ineligible during visit 1, prior to randomization.
Groups:
- Arm I (Protonated E-liquid, Unprotonated E-liquid): Visit 2: Patients sample protonated e-liquid
  Visit 3: Patients sample unprotonated e-liquid
- Arm II (Unprotonated E-liquid, Protonated E-liquid): Visit 2: Patients sample unprotonated e-liquid
  Visit 3: Patients sample protonated e-liquid
Period: Overall Study
Arm/Group | Arm I (Protonated E-liquid, Unprotonated E-liquid) | Arm II (Unprotonated E-liquid, Protonated E-liquid)
Started | 12 | 8
Sample Protonated E-liquid | 12 | 8
Sample Unprotonated E-liquid | 12 | 8
Completed | 12 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Protonated E-liquid, Unprotonated E-liquid) | Arm II (Unprotonated E-liquid, Protonated E-liquid) | Total
Number analyzed (Participants) | 12 | 8 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.17 (7.91) | 31.50 (7.27) | 33.10 (7.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 5 | 4 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 6 | 18
  Middle Eastern | 0 | 1 | 1
  More than one race | 0 | 1 | 1
Years of regular e-cigarette use [Mean (Standard Deviation); unit: years] | 3.67 (2.84) | 4.13 (2.95) | 3.85 (2.81)

OUTCOME MEASURES:

1. Primary Outcome: PET/CT Imaging of the Head
Description: Evaluate effect of nicotine form (free-base vs nicotine salt base) on nicotine absorption and distribution in the brain with total absorbed dose (TAD) of [11C]nicotine.
Time Frame: 1.5 hours
Population: Scan data from 3 participants was insufficient for calculating TAD and are not included in the statistics presented here, these participants were used for protocol optimizations.
Measure: Mean (Standard Deviation); unit: %TAD/kg
Units Other Than Participants: PET Scans
Groups:
- Protonated E-liquid: Patients sample protonated e-liquid
- Unprotonated E-liquid: Patients sample unprotonated e-liquid
Arm/Group | Protonated E-liquid | Unprotonated E-liquid
Number analyzed (Participants) | 17 | 17
Number analyzed (PET Scans) | 34 | 34
%TAD/kg | 2.81 (0.92) | 2.40 (0.62)

2. Primary Outcome: PET/CT Imaging of the Chest
Description: Evaluate effect of nicotine form (free-base vs nicotine salt base) on nicotine absorption and distribution in the respiratory tract with total absorbed dose (TAD) of [11C]nicotine.
Time Frame: 1.5 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: %TAD/kg
Units Other Than Participants: PET Scans
Arm/Group | Protonated E-liquid | Unprotonated E-liquid
Number analyzed (Participants) | 17 | 17
Number analyzed (PET Scans) | 34 | 34
%TAD/kg
  Upper Respiratory Tract | 6.18 (2.17) | 11.62 (3.17)
  Lower Respiratory Tract | 10.35 (3.49) | 5.53 (0.81)

3. Primary Outcome: Puff Volume (mL)
Description: Puffing topography data was captured by the study e-cigarette to determine the puff volume.
Time Frame: approx. 30 minutes
Population: Puffing topography was not able to be recorded for 2 participants while sampling the Protonated e-liquid and 1 participant while sampling the Unprotonated e-liquid.
Measure: Mean (Standard Deviation); unit: mL
Units Other Than Participants: Puffs
Arm/Group | Protonated E-liquid | Unprotonated E-liquid
Number analyzed (Participants) | 18 | 19
Number analyzed (Puffs) | 35 | 36
mL | 79.35 (72.75) | 73.76 (70.82)

4. Primary Outcome: Puff Duration (s)
Description: Puffing topography data was captured by the study e-cigarette to determine the puff duration.
Time Frame: approx. 30 minutes
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: Puffs
Arm/Group | Protonated E-liquid | Unprotonated E-liquid
Number analyzed (Participants) | 18 | 19
Number analyzed (Puffs) | 35 | 36
seconds | 2.87 (1.43) | 2.82 (1.61)

5. Primary Outcome: Age of First Tobacco Use
Description: Age of first use will be assessed using the tobacco use history questionnaire.
Time Frame: approx. 5 minutes
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Arm I (Protonated E-liquid, Unprotonated E-liquid) | Arm II (Unprotonated E-liquid, Protonated E-liquid)
Number analyzed (Participants) | 12 | 8
years | 14.58 (2.02) | 14.63 (1.60)

6. Primary Outcome: Years of Tobacco Use
Description: Years of tobacco use will be assessed using the tobacco use history questionnaire.
Time Frame: approx. 5 minutes
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Arm I (Protonated E-liquid, Unprotonated E-liquid) | Arm II (Unprotonated E-liquid, Protonated E-liquid)
Number analyzed (Participants) | 12 | 8
years | 19.58 (8.85) | 16.88 (6.75)

7. Primary Outcome: Years of Regular Use of Nicotine/Tobacco Products
Description: Years of regular use of nicotine/tobacco products will be assessed using the tobacco history questionnaire
Time Frame: approx. 5 minutes
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Arm I (Protonated E-liquid, Unprotonated E-liquid) | Arm II (Unprotonated E-liquid, Protonated E-liquid)
Number analyzed (Participants) | 12 | 8
years | 16.83 (8.99) | 15.13 (6.90)

8. Primary Outcome: Past 30 Day Use of Nicotine/Tobacco Products
Description: Days used in the past 30 days of nicotine/tobacco products including cigars, cigarillos, little cigars, pipe tobacco, chewing tobacco, snuff, snus, EC/vape/mod/APV/e-hookah, and hookah tobacco.
Time Frame: approx. 5 minutes
Population: 2 participants in Arm I declined to provide a response for the number of days they have used cigarettes in the past 30 days.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm I (Protonated E-liquid, Unprotonated E-liquid) | Arm II (Unprotonated E-liquid, Protonated E-liquid)
Number analyzed (Participants) | 12 | 8
days
  Cigarettes: number analyzed (Participants) | 10 | 8
  Cigarettes | 0 (0) | 0.75 (2.12)
  Pipes | 0 (0) | 0 (0)
  Cigars | 0 (0) | 0 (0)
  Cigarillos | 0 (0) | 0 (0)
  Little Cigars | 0 (0) | 0 (0)
  e-cigarettes | 29.83 (0.58) | 30.00 (0)
  Smokeless Tobacco | 0 (0) | 0 (0)
  Snus | 0 (0) | 0 (0)
  Hookah | 0.17 (0.58) | 0 (0)

9. Primary Outcome: Modified Cigarette Evaluation Questionnaire (mCEQ)
Description: 12-item modified Cigarette Evaluation Questionnaire (mCEQ) completed following e-cigarette self-administration to assess subjective responses. The 12-item mCEQ includes five subscales: Smoking Satisfaction, Psychological Reward, Aversion, Enjoyment of Respiratory Tract Sensations, and Craving Reduction, with items rated from 0 (not at all) to 6 (extremely likely). Scores for each subscale are calculated as the mean of the individual item responses or the single item. Higher scores indicate greater intensity on that scale.
Time Frame: approx. 5 minutes
Population: mCEQ was only evaluated during the second study visit
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Protonated E-liquid | Unprotonated E-liquid
Number analyzed (Participants) | 12 | 8
Score on a scale
  Satisfaction | 2.28 (1.31) | 1.42 (0.92)
  Psychological Reward | 2.17 (1.27) | 1.38 (0.93)
  Aversion | 0.88 (1.05) | 0.94 (1.47)
  Enjoyment of Respiratory Tract Sensations | 2.42 (1.31) | 1.25 (1.16)
  Craving Reduction | 3.67 (2.10) | 3.25 (1.83)

10. Primary Outcome: Drug Effects Liking Questionnaire (DEQ)
Description: An adapted version of the Drug Effects/Liking Questionnaire will assess the desire and liking of the study products. Five visual analog scale items ranging from 0 (not at all) to 100 (extremely) assessed wanting to vape the product again, liking the product, enjoying the product, finding the product pleasurable and satisfying. Higher scores indicate greater liking.
Time Frame: approx. 5 minutes
Population: The drug effects liking questionnaire was only administered during the second study visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Protonated E-liquid | Unprotonated E-liquid
Number analyzed (Participants) | 12 | 8
units on a scale
  Want | 60.08 (29.44) | 42.88 (26.69)
  Like | 51.25 (32.76) | 32.50 (25.93)
  Enjoy | 57.25 (30.63) | 31.88 (26.38)
  Pleasurable | 56.08 (32.42) | 29.13 (26.94)
  Satisfying | 60.33 (32.66) | 35.63 (28.54)

11. Primary Outcome: Modified Tiffany-Drobes Questionnaire of Smoking Urges: Brief Form (QSU)
Description: Urges/craving will be measured using a modified version of the Tiffany-Drobes Questionnaire of Smoking Urges: Brief Form. This is a 10-item measure where participants rate e-cigarette smoking-related items (All I want right now is an e-cigarette) on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). Similar to previous studies, we will collapse the items into two previously identified factors (Factor 1: strong desire and intention to smoke an e-cigarette; Factor 2: anticipation of relief from withdrawal symptoms). Scores are calculated by summing the items and range from 5 to 35 with higher scores indicating greater craving to vape.
Time Frame: aprox. 5 minutes
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Protonated E-liquid | Unprotonated E-liquid
Number analyzed (Participants) | 20 | 20
Score on a scale
  Desire | 29.45 (6.83) | 30.15 (5.82)
  Relief | 16.35 (8.01) | 17.40 (9.38)

12. Primary Outcome: Minnesota Nicotine Withdrawal Scale
Description: Nicotine withdrawal will be assessed using the empirically validated 15-item version of the Minnesota Nicotine Withdrawal Scale (MNWS). Items were rated on a 5-point scale from 0 (none) to 4 (severe). This measure assesses smoking craving, anger/irritability, anxiety, depressed mood, restlessness/difficulty concentrating, increased appetite, sleep problems, and somatic symptoms (nausea, constipation, sore throat, dizziness, coughing). MNWS is the sum of 8 items with scores ranging from 0 to 32 and MNWS Craving is a single item with scores ranging from 0 to 4, higher scores indicate a greater craving.
Time Frame: approx. 5 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Protonated E-liquid | Unprotonated E-liquid
Number analyzed (Participants) | 20 | 20
score on a scale
  MNWS | 9.50 (7.38) | 9.10 (6.32)
  MNWS Craving | 2.60 (0.94) | 2.70 (1.17)

13. Primary Outcome: Exhaled Breath Carbon Monoxide (CO)
Description: Exhaled breath carbon monoxide was collected before each scan with a handheld electrochemical device.
Time Frame: approx. 5 minutes
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Protonated E-liquid | Unprotonated E-liquid
Number analyzed (Participants) | 20 | 20
ppm | 2.45 (1.79) | 2.80 (2.31)

ADVERSE EVENTS:
Time Frame: Over 3 study visits, up to 3 months
Arm/Group | Protonated E-liquid | Unprotonated E-liquid
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 2/20 | 0/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Protonated E-liquid (N=20) | Unprotonated E-liquid (N=20)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-26): https://cdn.clinicaltrials.gov/large-docs/86/NCT05455086/Prot_SAP_000.pdf